CLINICAL TRIAL: NCT04408079
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance, Efficacy and Pharmacokinetics of TQB3558 Tablets
Brief Title: A Study to Evaluate the Tolerance, Efficacy and Pharmacokinetics of TQB3558 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3558-Ⅰ-01
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3558 Tablets (Experimental): TQB3558 tablets administered orally once. Then TQB3558 tablet administered orally, once daily in 28-day cycle after 4 days of first administration.
  Interventions: Drug: TQB3558

INTERVENTIONS:
Drug: TQB3558 — TQB3558 is a kinase inhibitor of the TRK protein family.

SUMMARY:
This is a study to evaluate the maximum tolerated dose (MTD) , occurrence of all adverse events (AE) and serious adverse events (SAE) , pharmacokinetic parameters and antitumor effect of TQB3558 tablets in Chinese adult patients with advanced solid tumors .The study is divided into phase Ia and phase Ib. Phase Ia: dose escalation period, to evaluate the safety and tolerability of TQB3558 tablets, determine MTD; Phase Ib: effectiveness exploration period, to expand the safe and effective dose group, recommend appropriate dosage and method for subsequent clinical research.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed advanced malignant solid tumors, without conventional treatment methods or fail or relapse after treatment.

  2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; Life expectancy ≥12 weeks.

  3. Has at least one measurable lesion (based on RECIST 1.1) or bone metastases. 4. Adequate organ system function. 5. Patients need to adopt effective methods of contraception. 6. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has received TRK inhibitors. 2. Has participated in any other clinical trials, or used other anti-cancer drugs, or received major surgical operations within 4 weeks before first administration.

  3. Has received local radiotherapy within 7 days or bone marrow radiotherapy within 4 weeks before the first administration.

  4. Has other malignant tumors in 2 years, except for cured or locally curable cancers.

  5. Has known spinal cord compression and cancerous meningitis. 6. Has interstitial lung disease, drug-induced interstitial lung disease, history of radiation lung disease requiring steroid therapy.

  7. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage.

  8. Obvious cardiovascular diseases. 9. Has a history of autoimmune disease, immunodeficiency. 10. Lactating women. 11. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 28 days
  MTD was defined as the dose in which more than 2 of up to 6 patients developed a DLT.
Adverse events (AE) and serious adverse events (SAE) | Baseline up to 28 days
  The occurrence of all adverse events (AE) and serious adverse events (SAE).
Overall response rate (ORR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Tmax | 15minutes, 30minutes, 1hour, 2hour, 4hour, 6hour, 8hour,10hour, 24hour, 48hour post-dose on day 1 and day 11; 30minutes pre-dose on day 1, day 5, day 7,day 8 ,day 9 and day 11.
  To characterize the pharmacokinetics of TQB3558 by assessment of time to reach maximum plasma concentration.
Cmax | 15minutes, 30minutes, 1hour, 2hour, 4hour, 6hour, 8hour,10hour, 24hour, 48hour post-dose on day 1 and day 11; 30minutes pre-dose on day 1, day 5, day 7,day 8 ,day 9 and day 11.
  Cmax is the maximum plasma concentration of TQB3558 or metabolite(s).
AUC0-t | 15minutes, 30minutes, 1hour, 2hour, 4hour, 6hour, 8hour,10hour, 24hour, 48hour post-dose on day 1 and day 11; 30minutes pre-dose on day 1, day 5, day 7,day 8 ,day 9 and day 11.
  To characterize the pharmacokinetics of TQB3558 by assessment of area under the plasma concentration time curve from zero to infinity.
CL/f | 15minutes, 30minutes, 1hour, 2hour, 4hour, 6hour, 8hour,10hour, 24hour, 48hour post-dose on day 1 and day 11; 30minutes pre-dose on day 1, day 5, day 7,day 8 ,day 9 and day 11.
  CL/f is total clearance rate for TQB3558.
Disease control rate（DCR） | up to 96 weeks
  Percentage of participants achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China